CLINICAL TRIAL: NCT00470691
Title: Comparison of Dorsal Plaster Splint and Circular Plaster Cast for Colles' Fractures
Brief Title: Dorsal Splint or Circular Cast for Colles' Fracture?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StOlavsH-ort-radius
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Colles' Fracture
MeSH Terms: conditions — Colles' Fracture | interventions — Casts, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- complete plaster cast (Experimental): reduction and a complete plaster cast,
  Interventions: Procedure: plaster cast
- dorsal plaster splint (Active Comparator): reduction and a dorsal plaster splint.
  Interventions: Procedure: dorsal splint

INTERVENTIONS:
Procedure: plaster cast — complete circular plaster cast
  Arms: complete plaster cast
Procedure: dorsal splint — dorsal plaster splint
  Arms: dorsal plaster splint

SUMMARY:
At our hospital, all Colles' fractures deemed suitable for conservative treatment are reduced and immobilised with a plaster of Paris dorsal splint which is converted to a complete cast after 10 days. According to individual factors such as age, general health and radiological results after 10 days, some patients with severe redisplacement are readmitted to hospital for surgery.

The main purpose of this study is to determine whether, during the first 10 days of immobilisation, a complete plaster cast or a dorsal plaster splint best retains the alignment of a reduced Colles' fracture. In addition, we aim to compare the complication rates of the two methods.

ELIGIBILITY:
Inclusion Criteria:

* women 50 years and older
* Colles' fracture due to low energy trauma

Exclusion Criteria:

* high energy trauma
* age under 50 years
* dementia

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2004-06; Primary Completion 2008-01 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
redisplacement | 10 days
  dorsal angulation, radial tilt and radial shortening - radiographs

SECONDARY OUTCOMES:
pain | 10 days
  pain during past 24h on a VAS
number of analgesic tablets | 10 days
  number of analgesic tablets taken during the 10 days after reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Vilh Finsen, MD, PhD, Study Chair — Dept of orthopaedic Surgery, St Olavs Hospital
Locations (1):
- St. Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Wik TS, Aurstad AT, Finsen V. Colles' fracture: dorsal splint or complete cast during the first 10 days? Injury. 2009 Apr;40(4):400-4. doi: 10.1016/j.injury.2008.08.044. Epub 2009 Feb 4. PMID 19195651